CLINICAL TRIAL: NCT01433302
Title: Determination of the Effect of Lymphatico-venous Bypass Surgery on Inflammatory Responses and Tissue Fibrosis
Brief Title: Inflammatory Response and Tissue Fibrosis/ Lymphatico-venous Bypass
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2011-0455; BC103691 (Other: Department of Defense)
Record Dates: First submitted 2011-09-08; First posted 2011-09-13 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer; Genitourinary Cancer; Malignant Female Reproductive System Neoplasm; Melanoma; Sarcoma
Keywords: Breast cancer; Genitourinary cancer; Gynecological cancer; Malignant Female Reproductive System Neoplasm; Melanoma; Sarcoma; Inflammatory Response; Inflammatory proteins; Tissue Fibrosis; Lymphatico-venous Bypass Surgery; Punch biopsy; Lab collections; Th2 immune phenotype; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Urogenital Neoplasms; Melanoma; Sarcoma; Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Punch Biopsy
  Interventions: Procedure: Punch Biopsy

INTERVENTIONS:
Procedure: Punch Biopsy — 5 mm punch biopsy specimens from the affected, lymphedematous limb will be obtained just prior to lymphatico-venular bypass and six (6) months after lymphatico-venular bypass. Punch biopsies will be obtained from the radial (lateral) aspect of the upper arm approximately 10cm above the olecranon process. Biopsy specimens will be collected from the contralateral (normal) arm at the exact same location.

SUMMARY:
The goal of this clinical research study is to measure the amount of inflammatory proteins inside the body before and after lymphatico-venular bypass surgery. This will help doctors learn if anti-fibrotic or anti-inflammatory drugs/treatments given with the surgery can improve how well the surgery works.

DETAILED DESCRIPTION:
If you choose to take part in this study, you will have 1 small piece of tissue (about the size of a pencil eraser) collected from the arm with the lymphedema and another small piece of tissue will be collected from the unaffected arm. A total of 4 samples will be collected by excisional biopsy (2 samples before the surgery and 2 more samples again 6 months after the surgery). To collect an excisional biopsy, the area of skin is numbed with anesthetic and a small cut is made to remove all or part of the affected tissue.

Blood (about 5 teaspoons each time) will also be drawn before the surgery and 1 more blood sample again 6 months after the surgery. If possible, the blood samples will be collected during already scheduled blood draws to avoid additional needle sticks.

The tissue and blood samples will be used for testing to evaluate the level of the tissue inflammation and to check for any build-up of excess tissue.

Length of Study:

After both tissue and blood samples have been collected, your participation in this study will be over.

This is an investigational study.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing lymphatico-venular bypass for lymphedema.
2. History of axillary lymph node dissection, sentinel lymph node biopsy or dissection.
3. A minimum of three (3) months post-op from any surgical interventions.
4. A minimum of six (6) months from the last dose of chemotherapy.
5. Patients with unilateral lymphedema.

Exclusion Criteria:

1. Active systemic infection or allergic reaction.
2. Active parasitic infection.
3. History of primary (congenital) lymphedema.
4. Metastatic cancer.
5. History of autoimmune disorders including lupus, rheumatoid arthritis, vasculitis, systemic sclerosis.
6. History of other fibroproliferative disorders including cirrhosis, pulmonary fibrosis, kidney fibrosis, systemic sclerosis, scleroderma.
7. Current treatment with steroids.
8. Concurrent secondary systemic cancer exclusive of cutaneous malignancies.
9. Treatment with myelosuppressive or stimulatory drugs within six (6) months of enrollment.
10. History of bone marrow transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UT MD Anderson Cancer Center patients, 18 years of age or older, undergoing lymphatico-venular bypass for stage II or greater lymphedema.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Th2 Cytokine Levels | 6 months
  5 mm punch biopsy specimens from the affected, lymphedematous limb will be obtained just prior to lymphatico-venular bypass and six (6) months after lymphatico-venular bypass. Punch biopsies will be obtained from the radial (lateral) aspect of the upper arm approximately 10cm above the olecranon process. Biopsy specimens will be collected from the contralateral (normal) arm at the exact same location.

CONTACTS AND LOCATIONS:
Overall Officials: David W. Chang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org